CLINICAL TRIAL: NCT02401919
Title: BASIC CARE REVISITED - Building the Evidence Base in Core Nursing Practice
Brief Title: Basic Care Revisited_Communication for Patient Participation
Acronym: BCR_C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 520002003
Record Dates: First submitted 2015-03-11; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Communication; Patient Participation
Keywords: Nursing; Hospital; Communication; Patient Participation; Individualised Care
MeSH Terms: conditions — Communication; Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tell-us Card Intervention (Experimental): Patients in the experimental arm will receive a Tell-us Card on a daily basis during their stay in the hospital. With this card patients are invited to state what is important to them for that day or before discharge from the ward.
  Interventions: Behavioral: Tell-us Card
- Care as usual (No Intervention): In the control arm, patients will receive care as usual.

INTERVENTIONS:
Behavioral: Tell-us Card — Patients will be invited on a daily basis, during their stay in the hospital, to state what is important for them at that moment or before discharge
  Arms: Tell-us Card Intervention

SUMMARY:
COMMUNICATION - Feasibility and effectiveness 'Tell-us Cards' in hospital patients

* Objective - To investigate the feasibility and effectiveness of 'Tell-us Cards' on patient participation in basic care in hospital settings.
* Design - Cluster randomised controlled early trial design (Phase 2B, MRC Framework). Patients of two surgical and two medical wards (n=140) will be included in this study. Before and after the introduction of the intervention, assessments will take place in patients and nurses at these wards.
* Intervention - The 'Tell-us card' is a tool to elicit patients preferences and needs in basic care. Patients are invited to write down their specific questions and concerns. The cards are handed out to patients admitted to the hospital (daily). Patients and informal caregivers are invited to use the cards to state their preferences. Nurses are instructed to use the cards as a tool in their dialogue with the patient in making care plans, during ward rounds or for discharge information sessions.
* Comparison - Usual care
* Primary outcome - Patient perception of participation in care (Individualized Care Scale (ICS)
* Secondary - Use and content of the 'Tell-us Cards' actions taken by nurses as a consequence of what patients 'tell them' by means of the 'Tell-us Cards', Quality from the Patients' perspective (QPP), EQ-5D, and CQ satisfaction with communication & care in general

DETAILED DESCRIPTION:
Feasibility and effectiveness of the 'Tell-us Card' Communication Tool on hospital patients' perception of participation and quality of Care.

The use of 'Tell-us Cards' in basic care is an intervention facilitating communication for enhanced patient participation in basic care. The effectiveness of the card is tested by Jangland et al (18) in a population of patients admitted to the hospitals surgical wards. The use of the 'Tell-us Card' in this patient group resulted in significant improvements in patients abilities to participate in decisions about their nursing and medical care. In our study we will investigate feasibility and effectiveness of the 'Tell-us cards' in three different hospital settings; patients admitted to the hospitals' surgical and medical wards and in patients attending the hospitals' emergency department.

Aim: The aim of this study is to investigate feasibility and effectiveness of 'Tell-us Cards' for patients participation in basic care in three different hospital settings. Description of the Intervention: The 'Tell-us card' (18) is a tool to elicit patients preferences and needs in basic care. Patients are invited to write down their specific questions and concerns for the day or before discharge. 'Tell-us Cards' are handed out on a daily basis to patients admitted to the hospital. Patients and their informal caregivers are invited to use the 'Tell-us Card' to state their preferences in basic care during their stay in the hospital. Nurses are instructed to use the 'Tell-us card' as a tool in their dialogue with the patient in making care plans, during ward rounds or for discharge information sessions.

Design: Feasibility and effectiveness of the 'Tell-us Card' will be tested in a controlled early trial design (Phase 2B, MRC Framework). Trained nurses will be handing out the 'Tell-us Cards' on a daily basis to patients admitted to the hospital. Baseline assessments on patient participation will be conducted at all wards in patients and nurses before the introduction of the 'Tell-us Cards'. For the baseline assessment; Nurses and patients will be asked to fill in a questionnaire. The nurses receive a questionnaire in their postbox at the ward they are working on with an envelope for returning the questionnaire to the researcher. Patients will be asked to fill in a questionnaire one week after discharge from the hospital or one week after their visit to the emergency department. Assessment of effects of the intervention in patients at T1 will start 3 months after the introduction of the 'Tell-us Cards' at the intervention wards. Nurses will be asked to fill in the questionnaire again 6 months after they filled in the first questionnaire.

Patients & Settings: Hospital patients admitted to two surgical wards and two medical wards (n=4x35=140) will be included in this study. One surgical ward, one medical ward will be randomly assigned to the intervention and control group. Baseline and follow up assessments will take place in 35 patients per assessment per ward, resulting in 165 assessments at baseline, and 165 assessments at follow-up. Outcomes: Primary outcome is patient perception of participation in individualised care. For measurement of patient participation in patients admitted to the hospital we will use the Individualized Care Scale for patients (19-23). Secondary outcomes will comprehend perception of quality of care, assessed with the Quality from the Patients' perspective (QPP) questionnaire (24, 25) as well as the use and content of the 'Tell-us Cards' and the actions taken by nurses as a consequence of what patients 'tell them' by means of the 'Tell-us Cards'. As generic tools we will use the EQ-5D for measurement of Quality of life (www.euroqol.org) and one question from the consumer Quality index for patient experience (www.centrumklantervaringindezorg). Furthermore nurses' perception of individualised care will be assessed at baseline and follow-up with the Individualized Care Scale for nurses.

Analysis: Results are clustered at ward level. We will therefore perform a random effects regression model to estimate the effects on (surgical and medical) patients' perceptions of Individualised Care for the intervention versus the usual care group at follow-up. In this analysis, ward will be entered as random effect, and covariates in the model are patients' perceptions of Individualised Care at each ward at baseline.

Descriptive analysis will reveal the topics patients regard as most important during their stay. A thorough process analysis on the use of the Card en the actions taken as a consequence of the content of the cards, will give insight in feasibility and effectiveness of the 'Tell-us Card' in daily practice.

Timeline (21 months): 1-6 (6m):Preparation time; 7-9 (3m):T0-Baseline assessment; 10-12 (3m):'Tell-us Card' Intervention Introduction; 13-15 (3m):T1-assessment; 16-21 (6m):Data analysis and study reporting

ELIGIBILITY:
Inclusion Criteria:

* Speaking the Dutch language

Exclusion Criteria:

* No serious cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in the Individualised Care Scale score | For patients at baseline and 4 months after the start start of the implementation proces
  Patients will receive a questionnaire at discharge
Change in Quality of Care Scale score | At baseline and 4 months after the start start of the implementation proces
  Patients will receive a questionnaire at discharge

SECONDARY OUTCOMES:
Process analysis 'Content of the Tell-us Card' | 3 months (after finalising implementation)
  The content of what patients report to be important for them during their stay or before discharge will be inventorized
Process analysis 'follow-up activities on content of Tell-us Card' | 3 months (after finalising implementation)
  The follow up activities by patients or nurses or other health professionals involved in care will be inventorized as well as the number of patients receiving the card, the number of patients indicating what is important for them during their stay or before discharge,

CONTACTS AND LOCATIONS:
Overall Officials: Ria Nijhuis-van der Sande, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud university medical center, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant

REFERENCES:
- [Background] Jangland E, Carlsson M, Lundgren E, Gunningberg L. The impact of an intervention to improve patient participation in a surgical care unit: a quasi-experimental study. Int J Nurs Stud. 2012 May;49(5):528-38. doi: 10.1016/j.ijnurstu.2011.10.024. Epub 2011 Nov 20. PMID 22104043
- [Background] Suhonen R, Schmidt LA, Katajisto J, Berg A, Idvall E, Kalafati M, Land L, Lemonidou C, Valimaki M, Leino-Kilpi H. Cross-cultural validity of the Individualised Care Scale - a Rasch model analysis. J Clin Nurs. 2013 Mar;22(5-6):648-60. doi: 10.1111/j.1365-2702.2012.04238.x. Epub 2012 Aug 9. PMID 22882146
- [Background] Suhonen R, Gustafsson ML, Katajisto J, Valimaki M, Leino-Kilpi H. Nurses' perceptions of individualized care. J Adv Nurs. 2010 May;66(5):1035-46. doi: 10.1111/j.1365-2648.2009.05256.x. Epub 2010 Mar 9. PMID 20337793